CLINICAL TRIAL: NCT00469703
Title: A Phase II, Open-Label, Single Center Pilot Study to Determine the Safety and Efficacy of THALOMID (Thalidomide) in Patients With Chronic Pancreatitis.
Brief Title: Safety and Efficacy Study of Thalomid in Patients With Chronic Pancreatitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated
Sponsor: Winthrop University Hospital (Other)
Collaborators: Celgene Corporation (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Chronic Pancreatitis
Record Dates: First submitted 2007-05-03; First posted 2007-05-04 (Estimated); Last update posted 2008-01-16 (Estimated); Status verified 2008-01

CONDITIONS: Chronic Pancreatitis
Keywords: Pancreatitis
MeSH Terms: conditions — Pancreatitis, Chronic; Pancreatitis | interventions — Thalidomide

INTERVENTIONS:
Drug: Thalidomide

SUMMARY:
The purpose of this study is to determine if Thalidomide (Thalomid) is effective in treating patients with chronic pancreatitis.

DETAILED DESCRIPTION:
Pancreatitis is an inflammation of the pancreas, a gland that lies behind the stomach. The inflammation may develop suddenly (acute pancreatitis) or over many years (chronic pancreatitis). The pancreas produces the hormones, insulin and glucagon to control metabolism. The hormones and enzymes flow from the pancreas through the pancreatic duct into the upper part of the small intestine.

Most chronic pancreatitis patients often experience chronic abdominal pain during the course of the disease. Thalidomide increased the production of interleukin-10 (IL-10), which is important in regulating intestinal inflammation. Thalidomide is approved by the Food and Drug Administration (FDA) for a leprosy skin condition, erythema nodosum lerosum (ENL), but not for the treatment of chronic pancreatitis. In this case it is considered experimental.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75, inclusive.
2. Female must be post menopausal (≥ 24 months without menses or surgically sterilized).
3. Able to comprehend English.
4. Chronic pancreatic pain lasting for more than 2 months.
5. History of chronic pancreatitis with pancreatic type pain confirmed by at least one of the following:

   * Histological confirmation
   * CT/MRI (including calcifications, dilated cuts, dilated MPD, and /or atrophy)
   * ERCP with Cambridge score of 2 or greater
6. Subject must score at least 4 cm on the VAS scale during the 1-2 week lead-in-period.
7. Patients must give written informed consent.
8. Patients must be willing and able to comply with the FDA-mandated S.T.E.P.S.® program.

Exclusion Criteria:

1. Female of child-bearing potential.
2. Unable to comprehend English.
3. Patients with diabetes requiring insulin.
4. Evidence of gallstones on screening ultrasonography.
5. Current alcohol abuse or addiction to opiate analgesics.
6. Patients with existing peripheral neuropathy.
7. Patients who are taking medications known to be associated with development of neuropathy: Amiodarone, hydralazine, perhexiline, vincristine, cisplatin, Metronidazole (Flagyl), Dapsone, Phenytoin and Disulfiram.
8. Patients who have pre-existing hypercoagulable state. Patients with a history of malignancy within the past 5 years, patients with a recent surgical procedure, patients with chronic immobilization causing blood stasis, patients with history of embolism or deep vein thrombosis, patients with extreme heart failure, and patients with a congenital disorder of the clotting cascade.
9. Patients with active alcoholic liver disease or elevated liver function >3Xs the upper limit of normal.
10. Patients will be withdrawn from the study at Visit 4 (Month 3) if pain score on VAS scale has not improved.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2005-08; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Safety and efficacy

SECONDARY OUTCOMES:
reduction of frequency of hospitalizations
quality of life
reduction of pain

CONTACTS AND LOCATIONS:
Overall Officials: James H Grendell, MD, Principal Investigator — Winthrop University Hospital